CLINICAL TRIAL: NCT03069105
Title: An Exploratory Study of Caregiver Burden Among Family Caregivers of Cancer Patients
Brief Title: An Exploratory Study of Caregiver Burden Among Family Caregivers of Patients With Cancer
Status: Completed | Type: Observational
Sponsor: Saint John's Cancer Institute (Other)
Responsible Party: Principal Investigator, Marlon Garzo Saria, Assistant Professor, Saint John's Cancer Institute
Other Study IDs: JWCI-16-1201
Record Dates: First submitted 2017-02-23; First posted 2017-03-03 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Caregivers; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Family caregivers: The sample for this study will consist of caregivers of patients with cancer. Eligible subjects who agrees to participate in the research study and sign the consent form will participate by completing paper and pencil or electronic questionnaires.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Participants will complete paper and pencil or electronic questionnaires at the cancer center or in the privacy of their own homes.

SUMMARY:
This study will look at caregiver burden and the coping behavior of caregivers of patients with cancer. Through this study, the investigators will identify the relationship between cognitive dysfunction (measured as a proxy rating by the caregiver), resilience, social support, cognitive appraisal, coping behavior, and caregiver burden, anxiety, and depression among family caregivers of patients with cancer.

DETAILED DESCRIPTION:
The goal of this study is to explore caregiver burden and the coping behavior of caregivers of patients with cancer. It has been documented that non-professional caregivers and long-term care providers to patients with cancer receive little preparation, information, or support to perform their vital role. Through this study, the investigators will identify the relationship between cognitive dysfunction, resilience, social support, cognitive appraisal, coping behavior, and caregiver burden, anxiety, and depression among family caregivers of patients with cancer. The findings of this study will direct future intervention studies to reduce caregiver burden and improve outcomes for the many individuals caring for family members with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Self-identified primary caregiver of patients with cancer
* Co-residence with the patient
* Providing a minimum of 4 hours of direct care for at least 3 days per week
* Able to speak, read, and understand English
* Willing to participate in completion of surveys

Exclusion Criteria:

* Professional or paid caregivers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample for this study will consist of caregivers of persons with cancer. A convenience sampling will be used to enroll eligible caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-04-28 (Actual)

PRIMARY OUTCOMES:
Changes in Caregiver Burden Score [Caregiver Reaction Assessment (CRA)] | 1 year
  Relation between caregiver burden subscale scores and caregiver resilience, social support, and coping

SECONDARY OUTCOMES:
Changes in Anxiety and Depression Score [Hospital Anxiety and Depression Scale (HADS)] | 1 year
  Relation between caregiver anxiety and depression score and caregiver resilience, social support, and coping

CONTACTS AND LOCATIONS:
Overall Officials: Santosh Kesari, MD PhD, Study Chair — Saint John's Cancer Institute; Marlon G Saria, PhD RN FAAN, Principal Investigator — John Wayne Cancer Institute at Providence Saint John's Health Center
Locations (4):
- United States (4):
  - Providence Saint Joseph Medical Center, Burbank, California
  - Providence Holy Cross Medical Center, Mission Hills, California
  - John Wayne Cancer Institute at Providence Saint John's Health Center, Santa Monica, California
  - EndBrainCancer Initiative/Chris Elliott Fund, Redmond, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saria MG, Nyamathi A, Phillips LR, Stanton AL, Evangelista L, Kesari S, Maliski S. The Hidden Morbidity of Cancer: Burden in Caregivers of Patients with Brain Metastases. Nurs Clin North Am. 2017 Mar;52(1):159-178. doi: 10.1016/j.cnur.2016.10.002. PMID 28189161
- [Background] Saria MG, Courchesne N, Evangelista L, Carter J, MacManus DA, Gorman MK, Nyamathi AM, Phillips LR, Piccioni D, Kesari S, Maliski S. Cognitive dysfunction in patients with brain metastases: influences on caregiver resilience and coping. Support Care Cancer. 2017 Apr;25(4):1247-1256. doi: 10.1007/s00520-016-3517-3. Epub 2016 Dec 5. PMID 27921222